CLINICAL TRIAL: NCT03044405
Title: Focused Assessed Echocardiography to Predict Fluid Responsiveness for Non-cardiac Hypotensive Spontaneously Breathing Patients After Major Abdominal Surgery
Brief Title: Focused Assessed Echocardiography to Predict Fluid Responsiveness
Acronym: fluidres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Asta Maculiene, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHO2
Record Dates: First submitted 2017-01-26; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypovolemia; Surgery; Hypotension
Keywords: fluid responsiveness; focused echocardiography; major surgery
MeSH Terms: conditions — Hypovolemia; Hypotension

STUDY DESIGN:
Intervention Model Description: Patients who had reduced arterial blood pressure up to 30% from the baseline after major abdominal surgery (gastric resection, gastrectomy, liver resection, pancreatic-duodenal resection, colorectal surgery) were included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Responders and non-responders (Other): Fluid challenge of 500 ml of crystalloids over 15 minutes is given. Positive fluid responsiveness is defined by an increase in stroke volume (SV) of at least 15% assessed by focused transthoracic echocardiography.
  Interventions: Diagnostic Test: Fluid challenge; Diagnostic Test: Focused transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Fluid challenge — Fluid bolus of 500 ml of crystalloids is given over 15 minutes. Positive fluid responsiveness is defined by an increase in SV of at least 15%.
Diagnostic Test: Focused transthoracic echocardiography — Focused transthoracic echocardiography is performed to assess expansion of stroke volume after fluid challenge. Also mitral E and A waves, left ventricle outflow tract velocity time integral (LVOT VTI) and its variability, inferior vena cava diameters during breathing cycles are measured.
  Other Names: extended hemodynamic monitoring

SUMMARY:
The aims of the study are:

1. To evaluate the feasibility of echocardiography monitoring in postoperative unit;
2. To assess diagnostic value of different focussed echocardiography parameters to define fluid responsiveness for non-cardiac hypotensive spontaneously breathing patients after major abdominal surgery.

DETAILED DESCRIPTION:
As there are different strategies of perioperative fluid management discussion which is the choice liberal or restrictive one occurs? Individualized infusion therapy should be the goal. The investigators hypothesize extended hemodynamic monitoring based on focused transthoracic echocardiography enable to differentiate the cause of hypotension more carefully and fluid overload will be avoided after major abdominal surgery.

The goals of the study are:

* To conduct one group of hypotensive patients after major abdominal surgery. To divide this group into responders and nonresponders after fluid challenge.
* To evaluate the feasibility of echocardiography monitoring in postoperative unit (having in mind such restrains as supine position, postoperative pain, bandages etc.)
* To compare the evaluation of fluid responsiveness by clinical signs and focused assessed echocardiography data.
* To identify the best focused echocardiography parameters for prognosis of fluid responsiveness.
* To determine if extended hemodynamic monitoring changes postoperative fluid management.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Patients who sign an agreement form to participate in the study.
* Patients undergoing major abdominal surgery.
* Hypotension

Exclusion Criteria:

* Younger than 18 years old.
* Known pregnancy.
* Unconscious patients or those who do not agree to participate in the study.
* Urgent surgery.
* Normal arterial blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
All hypotensive patients are divided into responders and non-responders according to increase of left ventricle outflow tract velocity time integral (LVOT VTI) after fluid challenge. | the first hour after the surgery
  Fluid challenge - fluid bolus of 500 ml of crystalloids which is given over 15 minutes. Positive fluid responsiveness is defined by an increase in stroke volume of at least 15%.
  Measurements are taken before and immediately after fluid challenge.

SECONDARY OUTCOMES:
The frequency of fluid responsiveness defined by clinical signs and focused transthoracic echocardiography data after fluid challenge is compared. | the first hour after the surgery
  Positive fluid responsiveness by clinical signs is defined as increase of arterial blood pressure more than 10mmHg after fluid challenge.
  Positive fluid responsiveness by focused transthoracic echocardiography data is defined as increase of LVOT VTI more than 15%.
Mitral E wave velocity (cm/s) is compared between responders and non-responders. | the first hour after the surgery
  Measurement is taken before the fluid challenge. The most reliable parameters to predict fluid responsiveness for non-cardiac hypotensive, spontaneously breathing patients after major abdominal surgery are assessed. The area under the curve (AUC) is defined to be clinically relevant if AUC is more than 0.7.
E/A ratio is compared between responders and non-responders. | the first hour after the surgery
  Measurement is taken before the fluid challenge. The most reliable parameters to predict fluid responsiveness for non-cardiac hypotensive, spontaneously breathing patients after major abdominal surgery are assessed. The area under the curve (AUC) is defined to be clinically relevant if AUC is more than 0.7.
Variability of LVOT VTI (%) during breathing cycles is compared between responders and non-responders. | the first hour after the surgery
  Measurement is taken before the fluid challenge. The most reliable parameters to predict fluid responsiveness for non-cardiac hypotensive, spontaneously breathing patients after major abdominal surgery are assessed. The area under the curve (AUC) is defined to be clinically relevant if AUC is more than 0.7.
Cardiac index (L/min/m2) is compared between responders and non-responders. | the first hour after the surgery
  Measurement is taken before the fluid challenge. The most reliable parameters to predict fluid responsiveness for non-cardiac hypotensive, spontaneously breathing patients after major abdominal surgery are assessed. The area under the curve (AUC) is defined to be clinically relevant if AUC is more than 0.7.
Variability of inferior vena cava (%) is compared between responders and non-responders. | the first hour after the surgery
  Measurement is taken before the fluid challenge.The most reliable parameters to predict fluid responsiveness for non-cardiac hypotensive, spontaneously breathing patients after major abdominal surgery are assessed. The area under the curve (AUC) is defined to be clinically relevant if AUC is more than 0.7.
The planed infusion therapy before and after evaluation by focused transthoracic echocardiography is compared in responders and non-responders. | the first 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Asta Maciuliene, M.D., Principal Investigator — Lithuanian University of Health Sciences; Andrius Macas, profesor, Study Chair — Lithuanian University of Health Sciences

IPD SHARING:
Plan to Share IPD: No